CLINICAL TRIAL: NCT04038801
Title: Clinical, Microbiological and Biochemical Effectiveness of Full-mouth Treatment Approaches in Severe Chronic Periodontitis: a Randomized Controlled Trial.
Brief Title: Full-mouth Treatment Approaches in Severe Chronic Periodontitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Beral Afacan, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMD
Record Dates: First submitted 2019-07-27; First posted 2019-07-31 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadrant-wise scaling and root planning (Q-SRP) (Active Comparator): Quadrant-wise scaling and root planing were performed over four visits at 1-weekly intervals using an assortment of manual periodontal curettes.
  Interventions: Procedure: Quadrant-wise scaling and root planning (Q-SRP)
- Full-mouth ultrasonic debridement (FMUD) (Experimental): Subgingival debridement were performed by a piezoceramic ultrasonic inserts in two visits of the same day.
  Interventions: Procedure: Full-mouth ultrasonic debridement (FMUD)
- Full-mouth disinfection (FMD) (Experimental): Subgingival debridement were performed by a piezoceramic ultrasonic inserts and an intensive regime of chlorhexidine in two visits of the same day.
  Interventions: Procedure: Full-mouth disinfection (FMD)

INTERVENTIONS:
Procedure: Quadrant-wise scaling and root planning (Q-SRP) — Quadrant-wise scaling and root planing were performed by assortment of manuel periodontal curettes over four visits at 1-weekly intervals.
  Arms: Quadrant-wise scaling and root planning (Q-SRP)
Procedure: Full-mouth ultrasonic debridement (FMUD) — Subgingival debridement were performed by a piezoceramic ultrasonic inserts in two visits of the same day.
  Arms: Full-mouth ultrasonic debridement (FMUD)
Procedure: Full-mouth disinfection (FMD) — Subgingival debridement were performed by a piezoceramic ultrasonic inserts and an intensive regime of chlorhexidine in two visits of the same day.
  Arms: Full-mouth disinfection (FMD)

SUMMARY:
This study aimed to compare the effects of full-mouth disinfection (FMD) and full-mouth ultrasonic debridement (FMUD) on clinical, microbiologic and biochemical parameters with conventional quadrant-wise scaling and root planning (Q-SRP) in patients with severe chronic periodontitis. 60 patients with severe chronic periodontitis were randomly allocated to three groups: FMD (n=20), FMUD (n=20) and Q-SRP (n=20). At baseline, gingival crevicular fluid (GCF) and subgingival plaque were collected and clinical periodontal parameters were recorded. Ultrasonic debridement was completed within 24 hours in FMD and FMUD groups. Chlorhexidine gluconate was used for FMD. Q-SRP was performed by hand instruments per quadrant at 1-week-intervals. Clinical parameters were recorded and samples were collected at 1, 3, 6 months after treatment. Real-time PCR was used for quantitative analysis of Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, Tannerella forsythia, Fusobacterium nucleatum and total bacteria count. Calprotectin, osteocalcin and cross-linked N-telopeptide of type I collagen (NTx) levels in GCF were analysed by enzyme-linked immunosorbent assay.

DETAILED DESCRIPTION:
Study population and clinical examination

60 consecutive severe chronic periodontitis patients were recruited for the study.

The whole mouth clinical periodontal examination included measurement of probing depth, clinical attachment level and plaque index at 6 sites per tooth, except the third molars The papillary bleeding index was recorded for the entire oral cavity. Clinical periodontal parameters were recorded at baseline and 1 month, 3 months and 6 months after treatments. Alveolar bone loss were assessed using an digital panoromic radiograph in each participant.

The diagnosis of severe chronic periodontitis was based on clinical and radiographic diagnostic criteria proposed by 1999 International Workshop for a Classification of Periodontal Diseases and Conditions. These individuals had a minimum of four non-adjacent teeth with sites with PD ≥6 mm and CAL ≥5 mm. They had also ≥50% alveolar bone loss in at least two quadrants that was commensurate with amount of plaque accumulation.

All clinical measurements, GCF and plaque sampling and also all treatments were performed by the same calibrated and trained investigator (B.A.) in a standardized manner (single-blinded trial).

Treatment

At the baseline visit, immediately before non-surgical periodontal treatment GCF and subgingival plaque samples were collected per patient and clinical periodontal measurements were recorded in all groups.

In the Q-SRP group, SRP were started with the upper right quadrant, and continued clockwise over four visits at 1-weekly intervals. SRP was performed using an assortment of manual periodontal curettes. The tooth surfaces were instrumented until it was visually and tactilely free of all deposits. Re-examinations were performed at 1, 3 and 6 months following the completion of the SRP in the lower right quadrant.

In the FMUD group, subgingival debridement were performed in upper jaw at the morning session and in lower jaw at the afternoon session. The procedure was completed in two visits (with 45 minutes interval) of the same day. All periodontal sites were debrided by a piezoceramic ultrasonic instrument with unmodified and modified inserts. Each tooth was instrumented till the root surface was visually and tactilely clean and smooth. Re-examinations were performed at 1, 3 and 6 months after the completion of full-mouth subgingival debridman.

In the FMD group, ultrasonic subgingival debridman was combined with an intensive antimicrobial regime with chlorhexidine. The dorsum of the tongue was brushed with a 1% chlorhexidine gel for 1 minute. The patients were instructed to rinse twice for 1 minute with 0.2% chlorhexidine solution. Each tonsil was sprayed four times with 0.2% chlorhexidine spray. Repeated subgingival irrigation with 1% chlorhexidine gel of all the pockets by a blunt needle. This subgingival application was repeated at day 8. For 14 days after the treatment, the patients were instructed to rinse twice daily for 1 min with 0.2% chlorhexidine solution and to spray the tonsils twice daily with a 0.2% chlorhexidine spray. Re-examinations were performed at 1, 3 and 6 months after 14 days washout period.

Standard oral hygiene instructions were given all patients immediately after the first session of Q-SRP group and the completion of the ultrasonic debridement in FMD and FMUD groups.

GCF sampling

GCF was sampled from the buccal aspects of two nonadjacent interproximal sites in single-rooted teeth with PD ≥6 mm, CAL ≥5 mm and visible signs of inflammation at baseline. Re-sampling was repeated at 1 month, 3 months and 6 months after treatment. Standardized filter paper strips were used for GCF sampling. The absorbed fluid volume was measured with a precalibrated electronic device. The paper strips were stored at -40◦C for further analysis.

Subgingival plaque sampling

After GCF collection, the subgingival plaque samples were collected from one site per quadrant with the deepest PD (≥5 mm) of single-rooted teeth at baseline and 1 month, 3 months and 6 months after treatment using two standardized no.30 sterile paper points. Pooled samples were stored at -40◦C for further analysis.

Measurement of calprotectin, osteocalcin, and NTx levels in GCF.

Two paper strips were pooled, placed in 300 microliter phosphatebuffered saline containing 0.05% polysorbate 20 and incubated for 20 minutes at room temperature on an orbital shaker. The fluid from the paper strips was recovered by centrifugation at 13 000 rpm for 5 minutes at +4◦C. Calprotectin, osteocalcin and NTx levels in GCF samples were measured by ELISA using commercial kits in line with the manufacturer's guidelines. Plates were measured at 450 nm with 650 nm as a reference wavelength by using an ELISA reader. Cytokine concentrations were calculated from the standard curve. GCF results were expressed as total amounts at two sites per sampling time.

Molecular detection of target bacteria in subgingival plaque.

The quantitative real-time PCR (qPCR) method was used for the quantitative detection of the selected periodontal pathogens in subgingival plaque. Total microbial DNA on paperpoints were extracted using High Pure PCR Template Preparation Kit according to the manufacturer's instructions. LightCycler FastStart DNA Master SYBR Green I Kit was used for the detection of target oligonucleotides according to the manufacturer's instructions. Real-time PCR protocols were constructed considering specific primer sets. Standard curves were constructed for the calculation of target oligonucleotides in the samples.

Statistical Analysis

Repeated measures analysis of variance (ANOVA) was used to detect intra- and intergroup differences in clinical, microbiological and biochemical parameters. Analysis of covariance was used for comparison of the improvements in parameters between the three treatment groups adjusting for the potential difference in the baseline data and Bonferroni test was performed post-hoc. The significance level was set at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥35 years
2. non-smokers
3. having at least 15 natural teeth.

Exclusion Criteria:

1. having any diagnosed medical disorder.
2. taken antibiotics, non-steroidal anti-inflammatory drugs, immunosuppressants, beta-blockers, calcium channel blockers within the past 6 months.
3. patients with a history of sensitivity to chlorhexidine.
4. nonsurgical/surgical periodontal treatment received in the past year
5. having a restorative and endodontic therapy requirement
6. having a removable partial denture and/or orthodontic appliances
7. current pregnancy or lactation.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2008-05-30 (Actual); Study Completion 2008-05-30 (Actual)

PRIMARY OUTCOMES:
GCF calprotectin | Change from baseline to 1, 3 and 6 months after treatment.
  Calprotectin (pg) levels in GCF.
GCF osteocalcin | Change from baseline to 1,3 and 6 months after treatment.
  Osteocalcin (ng) levels in GCF.
GCF NTx | Change from baseline to 1,3 and 6 months after treatment.
  NTx (nM BCE) levels in GCF.

REFERENCES:
- [Derived] Afacan B, Cinarcik S, Gurkan A, Ozdemir G, Ilhan HA, Vural C, Kose T, Emingil G. Full-mouth disinfection effects on gingival fluid calprotectin, osteocalcin, and N-telopeptide of Type I collagen in severe periodontitis. J Periodontol. 2020 May;91(5):638-650. doi: 10.1002/JPER.19-0445. Epub 2020 Mar 14. PMID 32023661